CLINICAL TRIAL: NCT03863405
Title: The Effect of Metformin on the Clinical Outcome of Patients With Rheumatoid Arthritis
Brief Title: Metformin Use in Rheumatoid Arthritis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Collaborators: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Mahmoud Mustafa Mahmoud Gharib, Principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 215
Record Dates: First submitted 2019-03-04; First posted 2019-03-05 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant
Masking Description: single blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin Group (Experimental): 850 mg metformin twice daily for six months in addition to standard therapy
  Interventions: Drug: Metformin; Drug: Conventional DMARDs
- Control Group (Active Comparator): placebo in addition to standard therapy for rheumatoid arthritis
  Interventions: Drug: Conventional DMARDs; Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Metformin — metformin 850 mg bid for RA patients with moderate to high disease activity provided by DAS-28 score greater than 3.2
  Arms: Metformin Group
Drug: Conventional DMARDs — methotrexate, leflunomide, hydroxychloroquine or sulfasalazine
Drug: Placebo Oral Tablet — oral tablet
  Arms: Control Group

SUMMARY:
Metformin has been used clinically for over 50 years, as a glucose lowering agent.

Direct and indirect anti-inflammatory effects of metformin have been reported in animal and clinical studies, and this effect is independent of its hypoglycemic effect.

Animal studies showed that metformin decreased serum C-reactive protein (CRP) level in atherogenic rabbits and decreased proinflammatory cytokines (interleukin (IL)-1β, IL-6 and tumor necrosis factor (TNF-α) in obese mice .

Moreover, metformin also suppressed osteoclastogenesis ; this may partially result from decreased expression of inflammatory cytokines that promote osteoclastogenesis in the arthritic joint.

The objective of this study is to evaluate the efficacy and safety of addition of metformin to standard disease modifying anti-rheumatic drugs (DMARDs) in patients with rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years (of both sexes) diagnosed with rheumatoid arthritis according to ACR / EULAR 2010 criteria .
* Patients with moderate to high disease activity (DAS - 28 . score greater than 3.2)
* Patients received the standard therapy (i.e. one or more conventional DMARDs) for at least three months.

Exclusion Criteria:

* Known hypersensitivity to metformin.
* Patients who have a prior diagnosis with diabetes mellitus.
* Patients receive metformin for any other indications.
* Patients with congestive heart failure.
* Patients with a history of myocardial infarction.
* Patients with severe anemia.
* Patients with active infections or other inflammatory diseases.
* Patients receiving biological therapy.
* Pregnancy or lactation.
* Patients with impaired liver functions.
* Patients with impaired kidney functions (serum creatinine concentrations ≥1.5 and ≥1.4 mg/dL in males and females respectively).
* Patients with malignancies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-01-09 (Actual); Primary Completion 2020-01-09 (Estimated); Study Completion 2020-01-09 (Estimated)

PRIMARY OUTCOMES:
disease activity scale in 28 joints ( DAS-28) | 6 months
  scale assessing severity of rheumatoid arthritis based on number of tender , swollen joints , ESR levels ,and patient self-assessment of his condition (global health assessment) . Whereas "28" describes the number of different joints including in the measurement :proximal interphalangeal joints (10 joints),metacarpophalangeal joints (10),wrists (2),elbows (2),shoulders (2),knees (2).
  DAS28 values range from 2 to 10 while higher values mean a higher disease activity. A DAS-28 value < 2.6 corresponds to remission,value between 2.6 and 3.2 corresponds to a low disease activity, value between 3.2 and 5.1 corresponds to a moderate disease activity, and DAS28 value >5.1 corresponds to a high disease activity.

SECONDARY OUTCOMES:
C reactive protein levels | 6 months
  blood samples will be withdrawn at baseline and after 3 and 6 months to evaluate serum levels of C reactive protein
The HAQ (Health Assessment Score) | 6 months
  HAQ-DI (Health Assessment Score- Disability index), in which patients are asked to rate their capacity to perform 20 activities of daily living (ADL). Scoring within each section is from 0 (without any difficulty) to 3 (unable to do). For each section the score given to that section is the worst score within the section, The Standard Disability Index (DI) calculated as the sum of the scores for various subscales divided by the number of subscales responded to, and results in a score between 0 and 3.Whereas scores can be interpreted as:
  From 0 to 1: mild difficulties to moderate disability, 2: moderate, 3: severe to very severe disability.
serum adiponectin level | 6-months
  blood samples will be withdrawn at baseline and after 3 and 6 months to evaluate serum adiponetin levels using ELISA kits
adverse effect incidence | 6 months
  adverse effect will be reported by patients or their caregivers and recorded by investigator

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Zahraa University Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No